CLINICAL TRIAL: NCT00283881
Title: Implicit Tactile Learning in Chronic Stroke Enhanced by Non-Invasive Brain Stimulation of the Somatosensory Cortex
Brief Title: Tactile Learning in Stroke Patients
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060080; 06-N-0080
Record Dates: First submitted 2006-01-29; First posted 2006-01-30 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-10-07

CONDITIONS: Stroke
Keywords: Haptic Skills; Implicit Tactile Learning; Functional Magnetic Resonance Imaging (fMRI); Transcranial Magnetic Stimulation (TMS); Transcranial Direct Current Stimulation (tDCS); Stroke; Healthy Volunteer; HV
MeSH Terms: conditions — Stroke

SUMMARY:
This study will determine if stimulation of the stroke-injured side of the brain combined with stimulation to the paralyzed hand can temporarily improve the sense of touch in stroke patients.

Healthy normal volunteers and people who have had a single stroke within 3 months of entering the study that affected one side of the brain may be eligible for this study. All participants must be between 18 and 90 years old and must be right-handed. Candidates are screened with a medical history, neurological examination and magnetic resonance imaging (MRI) of the brain if one has not been done within 1 year of entering the study.

Participants undergo the following tests and procedures during four 2-day sessions over about 6 weeks:

* Peripheral high-frequency stimulation: Small loudspeakers are taped to the fingertips and simple tactile pulses are passed through the skin. Stimulation may be sham or real.
* Transcranial direct current stimulation: Two small rubber electrodes are taped to the head - one above the eye and the other on the back of the head. A current is passed between the two electrodes. Stimulation may be sham or real.
* MRI: The subject lies in the scanner, a metal cylinder surrounded by a magnetic field, for about 40 minutes, lying still for up to 40 minutes at a time. An electrical stimulation is applied to the fingers of the right and left hand in separate sessions. Earplugs are worn to muffle the loud noises during the scanning. Functional MRI measures blood flow changes in the brain during the performance of specific tasks.
* Behavioral measurements:

  * Grating orientation task: The subject responds as quickly as possible to a touch stimulus to the finger by saying whether the direction of the stimulus is vertical or horizontal.
  * Haptic object recognition task: The subject is given five categories of unfamiliar objects in the shape of cubes. During the task, identical objects are hidden in a sack. With eyes closed, the subject is asked to identify and find the objects from the sack as quickly as possible.
  * Pegboard test: The subject is asked to place several pegs into a corresponding hole of a pegboard as soon as possible.
  * Tapping task: The subject is asked to tap a metal stick on a metal plate as quickly as possible for 1 minute.
* Paired-pulse transcranial magnetic stimulation: This test measures changes in brain activity. A wire coil is held on the scalp and a brief electrical current is passed through the coil, creating a magnetic pulse that stimulates the brain. The subject hears a click and may fee a pulling sensation on the skin under the coil, and there may be a twitch in the muscles of the face, arm or leg. Subjects may be asked to tense certain muscles slightly or perform other simple actions.
* Paired-pulse somatosensory evoked potential mapping: This test measures brain activity in another brain area. The subject is seated in a chair with eyes closed. One electrode is placed above the eye and two others are placed on the back of the head. A short electrical stimulus is applied to a nerve in the wrist and brain activity is recorded while the stimulus is applied.
* Surface electromyography: This test measures the electrical activity of muscles. Electrodes are filed with a conductive gel and taped to the skin.
* Visual analog and mood scale: Subjects complete questionnaires about their attention, fatigue and mood.

DETAILED DESCRIPTION:
Chronic stroke is often accompanied by tactile impairments that contribute to long-term disability in activities of daily living. While new rehabilitative interventions recently became available in the motor domain by using transcranial direct current stimulation (tDCS), there is no generally accepted treatment for tactile impairments after chronic stroke. Previous studies in healthy volunteers demonstrated that tactile acuity and haptic skills can be improved by applying a passive learning protocol to the fingertip (peripheral high-frequency stimulation, pHFS). Based on these findings, the purpose of this protocol is to enhance the beneficial effect of pHFS on implicit tactile and haptic learning in chronic stroke patients by a combined application of pHFS with tDCS (pHFS+tDCS) applied to the somatosensory cortex of the affected hemisphere. This approach might identify novel strategies to enhance functional recovery after stroke and might provide deeper insight into mechanistic information on the neural substrates involved in these behavioral gains. Primary outcome measures will be performance in a tactile grating orientation discrimination task (GOT) and in a haptic object recognition task. In order to obtain descriptive preliminary information on the relation between sensory improvements and motor deficits in chronic stroke patients, secondary outcome measures will be fine motor tasks such as a tapping task and a pegboard test (PBT) that require manual dexterity, handeye coordination, steadiness, and perceptual motor skills. To identify the operating mechanisms underlying hypothesized performance improvements after pHFS+tDCS, we will use paired-pulse protocols to evaluate changes in cortical excitability as well as fMRI in a subset of patients to identify cortical map reorganization in primary (SI) and secondary (SII) somatosensory cortex as well as in primary motor cortex (MI). Healthy volunteers will be tested (a) since there are no data available on performance of the haptic task in healthy subjects, (b) to obtain descriptive information on the influence of our interventions on this task for hypothesis generation purposes in our future investigations, and (c) because sensorimotor performance in the non-paretic hand of stroke patients is often not normal and therefore a poor sole control for performance of the paretic hand. Studies in chronic stroke patients will help address the main experimental hypothesis.

ELIGIBILITY:
* INCLUSION CRITERIA:

We will include left- and right-handed stroke patients, aged 18-90 years, with thromboembolic or hemorrhagic hemispheric lesions at least 3 months after the stroke. We will choose patients who initially had a severe motor paresis (below MRC grade 2), and subsequently recovered to the point that they have a residual motor deficit but can perform the required tasks. Moreover, only chronic stroke patients with moderate tactile deficits (defined by absolute touch thresholds below 4 N using von Frey filaments) who are able to differentiate the alignment of a grating dome (either orthogonal or parallel to the index finger) of at least 5 mm grooves that is applied on the fingertip will be included in the protocol.

Assessment of the initial functional state will be taken either from patient reports or medical records. Right-handed healthy volunteers, aged 18-90 years, should be able to concentrate on the required tasks. Handedness will be assessed by the Edinburgh inventory scale as well as the hand dominance test (HDT). We will additionally perform a pregnancy test for women of child-bearing potential. All experimental sessions will be on outpatient basis.

EXCLUSION CRITERIA:

Chronic stroke patients will be not be eligible for the study if they:

* are unable to perform the behavioral tasks,
* have a sensory neglect,
* have had more than one clinical stroke,
* have both sides of the brain affected,
* have had a stroke in the cerebellum or brainstem,
* have a history of alcohol or drug abuse or severe language disturbances or serious cognitive deficits,
* have uncontrolled medical problems, such as heart, lung or kidney disease, epilepsy or diabetes mellitus,
* have severe tactile deficits (defined by Frey filaments exerting a force of 4 N to the distal pad of the finger on the paretic and non-paretic hand),
* are pregnant,
* have a cardiac pacemaker, intracardiac lines, implanted medication pumps, neural stimulators, metal in the cranium, with the exception of dental braces in the mouth.

Exclusion criteria for healthy volunteers:

Healthy volunteers will not be eligible for the study if they:

* are unable to perform the tasks,
* have a history of alcohol or drug abuse or severe language disturbances or serious cognitive deficits,
* have uncontrolled medical problems, such as heart, lung or kidney disease, epilepsy or diabetes mellitus,
* have severe tactile deficits (defined by Frey filaments exerting a force of 4 N to the distal pad of the finger),
* are pregnant,
* have a cardiac pacemaker, intracardiac lines, implanted medication pumps, neural stimulators, metal in the cranium except in the mouth, dental braces.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2006-01-25; Primary Completion 2009-10-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hummel F, Celnik P, Giraux P, Floel A, Wu WH, Gerloff C, Cohen LG. Effects of non-invasive cortical stimulation on skilled motor function in chronic stroke. Brain. 2005 Mar;128(Pt 3):490-9. doi: 10.1093/brain/awh369. Epub 2005 Jan 5. PMID 15634731
- [Background] Vega A. Use of Purdue pegboard and finger tapping performance as a rapid screening test for brain damage. J Clin Psychol. 1969 Jul;25(3):255-8. doi: 10.1002/1097-4679(196907)25:33.0.co;2-v. No abstract available. PMID 5803245
- [Background] Mansur CG, Fregni F, Boggio PS, Riberto M, Gallucci-Neto J, Santos CM, Wagner T, Rigonatti SP, Marcolin MA, Pascual-Leone A. A sham stimulation-controlled trial of rTMS of the unaffected hemisphere in stroke patients. Neurology. 2005 May 24;64(10):1802-4. doi: 10.1212/01.WNL.0000161839.38079.92. PMID 15911819